CLINICAL TRIAL: NCT06580067
Title: A Pilot Study of Everyday Stress and Pain Intensity Reduction Intervention Via Tongues and Understanding Study in Adult Outpatients With Sickle Disease (ESPIRITU Study)
Brief Title: The Feasibility of the Pray Until Something Happens (PUSH) Intervention-OUTPATIENT
Acronym: ESPIRITU
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB202401269
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-01

CONDITIONS: Sickle Cell Disease; Stress; Pain
MeSH Terms: conditions — Anemia, Sickle Cell; Pain | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pray Until Something Happens (PUSH) video clip (Experimental): This intervention is a 30-minute petitionary prayer, named Pray Until Something Happens (PUSH) stress reduction intervention using a mobile smart device.
  Interventions: Behavioral: Pray Until Something Happens (PUSH); Behavioral: Self-monitoring
- Attention Control Group (Active Comparator): The second group will have access to the same internet-based application to track daily their stress and pain levels but will not be able to view our Pray Until Something Happens intervention.
  Interventions: Behavioral: Pray Until Something Happens (PUSH)

INTERVENTIONS:
Behavioral: Pray Until Something Happens (PUSH) — Self-monitoring of outcomes + alerts/reminders + use of PUSH
  Other Names: PUSH Prayer Fellowship
Behavioral: Self-monitoring — Self-monitoring of outcomes + alerts/reminder
  Arms: Pray Until Something Happens (PUSH) video clip

SUMMARY:
The goal of this research study is to reduce stress and improve sickle cell disease (SCD) pain control and sleep quality with less opioid use by determining the feasibility of an intervention with self-management combined intercessory and petitionary prayer, named Pray Until Something Happens (PUSH) stress reduction intervention using a mobile smart device. Currently, opioid analgesics are primarily used to treat SCD pain while self-managed behavioral modalities such as PUSH, are rarely used. Little is known about the effects or mechanisms of PUSH on pain, stress, and sleep symptoms in adults with SCD. Emerging evidence from the hypothalamic pituitary adrenal (HPA) axis theory offer insights for understanding the mechanisms. Adding PUSH as a supplement to analgesic therapies will address the dearth of self-management strategies for controlling pain in SCD. PUSH is a simple and cost-effective non-drug intervention that could reduce pain and stress in inpatients with SCD. GR is an intervention where inpatients with SCD are directed to listen to the audio recordings of the PUSH prayer session.

DETAILED DESCRIPTION:
The purpose of this research study is to see if a new computerized stress reduction program, called Pray Until Something Happens (PUSH) stress reduction intervention, can be used to teach people who have sickle cell disease (SCD) how to track their stress and pain daily and use guided audio-visual relaxation exercises to help them reduce their stress and pain. To obtain preliminary data for a larger randomized controlled trial, we propose to recruit 30 adult outpatients with SCD.

The investigators will stratify patients on worst pain intensity (<=5 and >5) and randomly assign 15 adults to Attention Control (Daily stress/pain tracking on Days 1-6) and 15 adults to Experimental (PUSH Prayer Fellowship on Day 1 and daily stress/pain tracking and PUSH intervention on Days 2-6) groups.

Immediate effects on pain, stress, and relaxation responses after the PUSH Prayer Fellowship will be examined. Patients will continue the trial for additional 6 days, with self-management on Days 2-6 and posttest on Day 7 while hospitalized to test short-term (7 days) effects of PUSH on outcomes (pain, stress, sleep quality, and opioid use).

During Days 2-6, the experimental group will participate in an audio/visual Zoom recorded prayer session that will be conducted specifically for each patient by the interventionist. Following the prayer session, the link to the recorded prayer is uploaded to the PAINReportIt program. Patients will access the recorded prayer session on Days 2-6. These patients will listen to the recorded PUSH prayer session at stress onset and as often as they desire. We will investigate mechanisms by which PUSH produces its effects in adult outpatients with SCD.

ELIGIBILITY:
Inclusion Criteria:

* Has SCD diagnosis;
* Reports pain 3 or greater in the previous 24 hours (0-10 scale)
* Speaks and reads English
* 18 years of age or older
* Uses opioid analgesics on "as needed" or "continuous" basis
* Allows healing prayers to be offered for them in the name of Jesus Christ

Exclusion Criteria:

* Legally blind
* Physically or cognitively unable to complete study measures

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Current Pain | Immediate (Day 1 baseline) and Days 2-7
  Patient-Reported Outcomes Measurement Information System (PROMIS) Pain intensity scale: A 3-item scale that asks patients to report their pain now, worst, and average on a scale of 1 to 5 where 1 is "had no pain" and 5 is "very severe." We will estimate intervention effects using regression analysis.
Average pain intensity | Short-term (Day 7)
  A 3-item scale that asks patients to report their current, least, and worst pain intensity today, on a scale of 0 to 10, where 0 is "no pain" and 10 is "pain as bad as it could be." We will average the three scores to create an average pain intensity score. We will estimate intervention effects using linear regression.

SECONDARY OUTCOMES:
Current stress | Immediate (Day 1 baseline) and Days 2-7
  Stress intensity scale: A 3-item scale that asks patients to report their current, least, and worst stress intensity today, on a scale of 0 to 10, where 0 is "no stress" and 10 is "stress as bad as it could be." We will estimate intervention effects using linear regression.
Average stress intensity | Short-term (Day 7)
  Stress intensity scale: A 3-item scale that asks patients to report their current, least, and worst stress intensity today, on a scale of 0 to 10, where 0 is "no stress" and 10 is "stress as bad as it could be." We will average the three scores to create an average stress intensity score. We will estimate intervention effects using linear regression.
Sleep quality | Immediate (Day 1 baseline) and Short-term (Day 7)
  Sleep quality scale: A self-administered questionnaire that incorporates a discretizing VAS. The questionnaire instructions direct the respondent to rate the overall quality of sleep over a 7-day recall period on a discretizing VAS, whereby the respondent marks an integer score from 0 to 10, according to the following five categories: 0 = terrible, 1-3 = poor, 4-6 = fair, 7-9 = good, and 10 = excellent. When rating their sleep quality, respondents are instructed to consider the following core components of sleep quality: how many hours of sleep they had, how easily they fell asleep, how often they woke up during the night (except to go to the bathroom), how often they woke up earlier than they had to in the morning, and how refreshing their sleep was.
Opioid use | Immediate (Day 1 baseline) and Short-term (Day 7)

OTHER OUTCOMES:
Perceived stress | Immediate (baseline)
  Perceived Stress Questionnaire: A 30-item questionnaire that measures perceived stress in the last two weeks. An overall perceived stress index (PSI) score for each scale is computed by subtracting 30 from the raw score and dividing it by 90, yielding scores that range from 0 to 1. Higher scores indicate greater perceived stress recent. We will analyze data using linear regression.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam O Ezenwa,, PhD, RN, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States